CLINICAL TRIAL: NCT05668702
Title: A Comparison of Two Regions Used in Capillary Blood Glucose Test in Terms of Pain and Result Consistency
Brief Title: Blood Glucose Measurement in Terms Ofg Pain and Result Consistency
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melek Sahin (Other)
Responsible Party: Sponsor-Investigator, Melek Sahin, Principal Investigator, Muğla Sıtkı Koçman University
Organization: Muğla Sıtkı Koçman University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 05.04.2018 04/I
Record Dates: First submitted 2022-12-04; First posted 2022-12-30 (Actual); Last update posted 2022-12-30 (Actual); Status verified 2022-12

CONDITIONS: Glucose Test Site Bleeding
Keywords: pain; capillary blood sampling; fingertip; glucose
MeSH Terms: conditions — Pain | interventions — Cross-Over Studies

STUDY DESIGN:
Intervention Model Description: crossover design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- capillary blood glucose measurement (Experimental): the researcher took venous blood sample in a tube from each patient and according to the list of order determined via randomization scheme formed on the computer, the patients' glucose levels were measured by taking a capillary blood sample from the side of the middle fingertip and palm of the dominant hand with the glucometer. Before the study, the patient's pain assessment at the end of each measurement was carried out by a nurse who was trained by the researcher about the use of Visual Analog Scale.
  Interventions: Other: crossover design

INTERVENTIONS:
Other: crossover design — The researcher took venous blood sample in a tube from each patient and according to the list of order determined via randomization scheme formed on the computer, the patients' glucose levels were measured by taking a capillary blood sample from the side of the middle fingertip and palm of the dominant hand with the glucometer. Before the study, the patient's pain assessment at the end of each measurement was carried out by a nurse who was trained by the researcher about the use of Visual Analog Scale.
  Other Names: capillary blood glucose measurement; venous blood glucose measurement; pain assessment

SUMMARY:
Abstract Background: Capillary blood glucose measurement is one of the invasive procedures frequently used in clinics, hospitals and home.

Aim: To determine the consistency of pain and results between the palm and fingertip in obtaining blood sample with the intention of monitoring capillary blood glucose.

Design: This study is a crossover design designated. Settings: The research was carried out Diabetes Polyclinic Participants: One hundred thirty Type 2 diabetes patients who went to Diabetes Polyclinic Methods: The research was carried out with 130 Type 2 diabetes patients who went to Diabetes Polyclinic between August and November, 2018. During the data collection, the researcher took venous blood sample in a tube from each patient and according to the list of order determined via randomization scheme formed on the computer, the patients' glucose levels were measured by taking a capillary blood sample from the side of the middle fingertip and palm of the dominant hand with the glucometer. Before the study, the patient's pain assessment at the end of each measurement was carried out by a nurse who was trained by the researcher about the use of Visual Analog Scale.

Keywords: capillary blood sampling; fingertip; glucose; pain; palm

DETAILED DESCRIPTION:
Avoid duplicating information that will be entered elsewhere, such as Eligibility Criteria or Outcome Measures.

The data were collected by the researcher in the diabetes outpatient clinic where there is a sink for handwashing and a suitable area and equipment for blood collection. The researcher interviewed the patients who applied to the diabetes outpatient clinic, informed them about the study and obtained their written consents. After obtaining their written consents, the information of the patients was recorded in the Patient Identification Form. Then, the patients were informed about the use of the Visual Analog Scale. First, venous blood samples of the patients were collected into a tube by the researcher, and then their capillary blood samples were taken. A randomization scheme was created via the website https://www.randomizer.org/ in order to prevent bias during the evaluation of the pain felt due to drawing of capillary blood. According to this randomization order, patients were randomly assigned to one of the two groups. For capillary blood glucose measurement, two regions, fingertip and palm were used in every patient. In the first group, capillary blood glucose samples were taken first from the fingertip and then from the palm, and in the second group the capillary blood sample was first obtained from the palm and then the fingertip, and blood glucose measurements were made with the glucometer. The patient washed his/her hands with warm water and soap and dried them with a paper towel. Prior to capillary blood collection, the patient washed his/her hands with warm water, kept his hand below the level of the heart, waved downwards and gently massaged his/her fingertips in order to obtain appropriate amount of blood. The dominant hands of the patients were used to collect capillary blood samples. In order not to affect the research results, the same glucometer device was used for all capillary glucose measurements and a new 28G sterile lancet was used in each application. Between capillary blood glucose measurements, an average of 5 minutes was waited for pain assessment with VAS. In order to ensure the objectivity of the study, the nurse, who was trained by the researcher on the use of VAS before the study, evaluated the patient's pain at the end of each capillary blood glucose measurement by using VAS.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with Type 2 diabetes
* who fasted at least 8-12 hours before blood sampling,
* who were 18 years and older,
* volunteered to participate in the study

Exclusion Criteria:

* with mental problems,
* communication problems,
* vision problems,
* upper extremity amputations,
* peripheral neuropathy or decreased sensation in their hands,
* the ones in whom blood samples cannot be obtained from the arm veins due to plaster etc.,
* those who could not make the Visual Analog Scale (VAS) correctly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
venous blood samples | through study completion, an average of 1 year
  Venous blood samples of the patients were collected into a tube by the researcher.
Capillary blood glucose measurement | through study completion, an average of 1 year
  For capillary blood glucose measurement, two regions, fingertip and palm were used in every patient. The patient washed his/her hands with warm water and soap and dried them with a paper towel. Prior to capillary blood collection, the patient washed his/her hands with warm water, kept his hand below the level of the heart, waved downwards and gently massaged his/her fingertips in order to obtain appropriate amount of blood. The dominant hands of the patients were used to collect capillary blood samples. In order not to affect the research results, the same glucometer device was used for all capillary glucose measurements and a new 28G sterile lancet was used in each application.

SECONDARY OUTCOMES:
Visual Analog scale (VAS) | through study completion, an average of 1 year
  At the end of each capillary blood glucose measurement, the patient's pain was assessed using the VAS.
  Visual Analog scale (VAS) is a one-dimensional scale used to measure pain. The scale consists of a 100 mm long line, with the words "painlessness" on one end and "the most severe pain" on the other end. "0" denotes painlessness, "100" denotes the most severe pain. The scale can be used horizontally or vertically. In this study, VAS was used horizontally.

CONTACTS AND LOCATIONS:
Overall Officials: Eylem Ergün, RN, Study Director — +905302373049
Locations (1):
- Fethiye Goverment Hospital, Muğla, Fethiye, Turkey (Türkiye)

REFERENCES:
- [Background] Bijur PE, Silver W, Gallagher EJ. Reliability of the visual analog scale for measurement of acute pain. Acad Emerg Med. 2001 Dec;8(12):1153-7. doi: 10.1111/j.1553-2712.2001.tb01132.x. PMID 11733293
- [Background] Chlebowy DO, Hood S, LaJoie AS. Facilitators and barriers to self-management of type 2 diabetes among urban African American adults: focus group findings. Diabetes Educ. 2010 Nov-Dec;36(6):897-905. doi: 10.1177/0145721710385579. Epub 2010 Oct 25. PMID 20974906
- [Result] Anitha Pavithran A, Ramamoorthy L, Bs S, Murugesan R, Mj K. Comparison of Fingertip vs Palm Site Sampling on Pain Perception, and Variation in Capillary Blood Glucose Level among Patients with Diabetes Mellitus. J Caring Sci. 2020 Dec 1;9(4):182-187. doi: 10.34172/jcs.2020.028. eCollection 2020 Dec. PMID 33409161
- [Result] Anzalone P. Equivalence of earlobe site blood glucose testing with finger stick. Clin Nurs Res. 2008 Nov;17(4):251-61. doi: 10.1177/1054773808325050. PMID 18927259
- [Result] Bina DM, Anderson RL, Johnson ML, Bergenstal RM, Kendall DM. Clinical impact of prandial state, exercise, and site preparation on the equivalence of alternative-site blood glucose testing. Diabetes Care. 2003 Apr;26(4):981-5. doi: 10.2337/diacare.26.4.981. PMID 12663560
- [Result] Chan HY, Lau TS, Ho SY, Leung DY, Lee DT. The accuracy and acceptability of performing capillary blood glucose measurements at the earlobe. J Adv Nurs. 2016 Aug;72(8):1766-73. doi: 10.1111/jan.12944. Epub 2016 Mar 1. PMID 27380764
- [Result] Ergin E, Zaybak A. Effects of Different Methods Used to Take Blood Samples on Blood Glucose Measurements. Clin Nurs Res. 2022 Jan;31(1):29-38. doi: 10.1177/10547738211024782. Epub 2021 Jul 5. PMID 34218680
- [Result] Farmer L, Winfield C, Quatrara B, Letzkus L, Schenck P, Finneran P, Pollak D, McCaskill C, Nealy R, Conaway M. Does Site Matter? Comparing Accuracy and Patient Comfort of Blood Glucose Samples Taken From the Finger and Palm of the Perioperative Patient. J Perianesth Nurs. 2017 Dec;32(6):573-577. doi: 10.1016/j.jopan.2016.10.006. Epub 2017 Mar 22. PMID 29157763
- [Result] Guo J, Long Q, Li J, Wang X, Li Y, Jiang S, Sun M, Wiley J, Chen JL. Barriers and facilitators of self-monitoring of blood glucose engagement among women with gestational diabetes mellitus in China: A mixed-methods study. Midwifery. 2020 Nov;90:102797. doi: 10.1016/j.midw.2020.102797. Epub 2020 Jul 18. PMID 32755742